CLINICAL TRIAL: NCT03523403
Title: The Apple Study: Investigating the Effects of Whole Apple Consumption on Risk Factors for Chronic Metabolic Diseases in Overweight and Obese Adults
Brief Title: Obesity-related Health Benefits of Apples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government); Ontario Apple Growers (Unknown); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Lindsay Robinson, Associate Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UGuelph Apple Study; UofG2014-2028 (Other Grant/Funding Number: Ontario Ministry of Agriculture, Food and Rural Affairs); UofG2014-2028 (Other Grant/Funding Number: Ontario Apple Growers); REB#16JA013 (Other: Research Ethics Board, University of Guelph)
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obesity, Abdominal; Hyperlipidemias; Inflammation; Dysbiosis
Keywords: Obesity; Diet; Apples; Polyphenols; Soluble fibre; Blood lipids; Lipid digestion; Inflammation; Cytokines; Microbiota; Dysbiosis; Type 2 diabetes risk; Cardiovascular disease risk
MeSH Terms: conditions — Obesity, Abdominal; Hyperlipidemias; Inflammation; Dysbiosis; Obesity

STUDY DESIGN:
Intervention Model Description: All 60 participants will participate in the Chronic phase of the study, which will follow a randomized, controlled, parallel-arm design to investigate the effects of consuming 3 apples per day for 6 weeks. 30 of those 60 participants will also participate in the Acute phase of the study, which will follow a randomized, crossover design to investigate the effects of eating 3 apples in addition to a high-fat meal in one sitting.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Acute phase - intervention (Experimental): Participants will be asked to consume 3 whole apples and a high-fat meal (a mixture of commercially available whipping cream and milk, providing 1 g of fat per kg of body weight) within 30 minutes.
  Interventions: Other: Apples
- Acute phase - control (No Intervention): Participants will be asked to consume a high-fat meal (a mixture of commercially available whipping cream and milk, providing 1 g of fat per kg of body weight) within 30 minutes.
- Chronic phase - intervention group (Experimental): Participants will be asked to consume 3 whole apples per day for 6 weeks.
  Interventions: Other: Apples
- Chronic phase - control group (No Intervention): Participants will be asked to consume no apples per day for 6 weeks.

INTERVENTIONS:
Other: Apples — 3 whole Ontario-grown Gala apples
  Arms: Acute phase - intervention; Chronic phase - intervention group

SUMMARY:
Obesity is characterized by an underlying inflammatory state in which various inflammatory signaling molecules, termed cytokines, affect metabolic processes central to type 2 diabetes and cardiovascular disease; leading causes of disability and death in Ontario. Such obesity-associated inflammation is partly due to the movement of endotoxin (i.e. lipopolysaccharide (LPS), a cell wall component of Gram-negative bacteria) from the gut microbiota to the blood, resulting in elevated blood levels of LPS (a condition termed metabolic endotoxemia) that stimulates inflammation. Digestion of a high-fat meal increases blood LPS and is subsequently associated with inflammation and metabolic impairments. However, in this context, little is known about how the consumption of bioactive-rich foods, such as whole apples, can improve impaired inflammatory and metabolic responses in overweight and obese individuals. Apples are a key commodity to study given that they are Ontario's predominant fruit crop with the apple industry valued at approximately $400 million, they require little food preparation, and they are common in the diet year-round. There are some, but limited, reports of potential apple-induced health benefits related to reductions in inflammation and improved metabolic responses in lean/healthy individuals, but work in overweight and obese individuals is especially lacking. Thus, to address the gap in our understanding of how daily apple intake may improve the health consequences of obesity, we will conduct a randomized clinical trial in which overweight and obese adults will consume three Ontario-grown Gala apples (approximately 300 g) as part of their typical diet in one sitting (i.e. acute consumption) and/or daily for six weeks (i.e. chronic consumption). The Acute Apple Consumption phase of the study will follow a randomized crossover design in which participants' rate of gastric emptying, efficacy of dietary lipid digestion and absorption, and production of inflammatory cytokines and biomarkers of metabolism will be assessed before and after consuming a high-fat meal (designed to provide 1 g fat/kg body weight) with or without three apples in one sitting. The Chronic Apple Consumption phase of the study will follow a randomized, controlled, parallel-arm design in which participants' (fasting) production of inflammatory cytokines and biomarkers of metabolism, as well as their gut microbiota profile, will be assessed before and after consuming three apples (or no apples) daily for six weeks. We hypothesize that the consumption of three whole apples in one sitting and daily for six weeks will improve these parameters in overweight and obese individuals at risk of developing chronic metabolic diseases.

DETAILED DESCRIPTION:
This study will be conducted at the Human Nutraceutical Research Unit (HNRU) at the University of Guelph. The research will be carried out in accordance with the SOPs established by the HNRU, which formalize the Department of Human Health and Nutritional Sciences (HHNS) procedures to ensure that participant safety and comfort are consistently maintained throughout the research process and that university research standards are met. This study will be conducted in compliance with the Tri-Council Policy Statement 2.

Procedure 1 - Recruitment and screening:

A total of 60 participants will be recruited for this study. Interested individuals will complete a 15-minute phone screening questionnaire to assess initial eligibility. If eligible, a 30-minute in-person screening visit to the HNRU will be scheduled to confirm eligibility. Prior to initiation of the in-person screening visit activities, the appropriate consent form will be provided to and discussed with the potential participant, and will be signed. At the in-person screening visit, potential participants will be asked to:

* Complete an in-person screening questionnaire of health and lifestyle habits
* Have anthropometric measures taken, including body weight, height, waist circumference and blood pressure in private area by a study coordinator Next, the Acute and Chronic Apple Consumption phases of the study will be explained to eligible participants, and all questions will be answered. Finally, the appropriate consent form will be provided to and discussed with eligible participants, and will be signed.

Study design:

This study has two phases: Acute and Chronic Apple Consumption. The Acute phase will involve eating 3 whole Ontario-grown Gala apples in one sitting, whereas the Chronic phase will involve eating 3 apples or no apples daily for 6 weeks. All 60 eligible participants will be included in the Chronic phase, and will be invited to also participate in the Acute phase. There will be no consequences for refusing to participate in the Acute phase. 30 of the 60 participants will be included in the Acute phase on a "first come, first served" basis, and upon completion of the Acute phase, they will immediately start the Chronic phase of the study.

Relevant to Acute + Chronic phase participants:

The Acute phase will follow a randomized, cross-over study design. Participants who volunteer to also participate in the Acute phase will complete the Acute phase before starting the Chronic phase of the study. At least 7 days prior to the start of the Chronic phase activities, Acute phase participants will visit the HNRU for 1, 7-hour study visit (see below). Participants will eat 3 apples or no apples, plus consume a high-fat meal (whipping cream + milk, designed to provide 1 g fat/kg body weight) containing 1500 mg of acetaminophen within 30 minutes. Whether Acute phase participants consume 3 apples or no apples at their study visit 1 will be randomized. At least 7 days later, participants will start the Chronic phase of the study. At their study visit 2 participants will consume the opposite of what they consumed at study visit 1: either 3 apples or no apples, plus the high-fat meal containing 1500 mg of acetaminophen within 30 minutes. Acute phase participants' measurements taken at the study visit with no apple consumption (study visit 1 or 2) will serve as their baseline measurements for the Chronic phase.

The Chronic phase will follow a randomized, parallel group study design. Participants will be randomized to either the intervention or control group; the intervention group will eat 3 apples/day for 6 weeks, while the control group will eat no apples/day for 6 weeks. Participants will:

* Collect 6 fecal samples: 3 before and 3 at the end of the 6-week study
* Visit the HNRU for 2, 15-minute check-in visits (see below) at weeks 2 and 4 during the study
* Complete 3, 3-day food records: before and at the end of the 2-week run-in period, and within weeks 4 - 6 of the Chronic phase of the study
* Visit the HNRU for 1 hour at the end of week 6. Participants will:

  * Be asked to complete a questionnaire detailing information about their diet, lifestyle habits, and any health issues to report
  * Have anthropometric measures including body weight, height, waist/hip circumference and blood pressure taken in a private area by a trained study coordinator
  * Provide a fasting blood sample via venipuncture conducted by a HHNS-approved, qualified phlebotomist

Relevant to Chronic phase only participants:

The Chronic phase will follow a randomized, parallel group study design. Participants will be randomized to either the intervention or control group; the intervention group will eat 3 apples/day for 6 weeks, and the control group will eat no apples/day for 6 weeks. Participants will:

* Visit the HNRU for 2, 1-hour study visits, immediately before, and immediately after the 6-week study. Participants will:

  * Be asked to complete a questionnaire detailing information about their diet, lifestyle habits, and any health issues to report
  * Have anthropometric measures including body weight, height, waist/hip circumference and blood pressure taken in a private area by a trained study coordinator
  * Provide a fasting blood sample via venipuncture conducted by a HHNS-approved, qualified phlebotomist
* Collect 6 fecal samples: 3 before and 3 at the end of the 6-week study
* Visit the HNRU for 2, 15-minute check-in visits (see below) at weeks 2 and 4 during the study
* Complete 3, 3-day food records: before and at the end of the 2-week run-in period, and within weeks 4-6 of the Chronic phase of the study

Procedure 2 - Dietary guidelines:

All participants will be asked to follow our dietary guidelines outlining a low-polyphenol diet for 2 weeks prior to their first study visit, followed by a reduced polyphenol diet (less restricted than the 2-week run-in period) during the study.

Procedure 3 - Study visits:

Relevant to the Acute phase:

Participants will visit the HNRU after a 10-12 h overnight fast on day 1 after the 2-week run-in period. Participants will be asked to consume a standardized evening meal consisting of a frozen vegetable lasagna, granola bar, pudding cup, and juice box prior to the 10-12 h overnight fast, and to avoid over-the-counter acetaminophen-containing products for 24 h, and alcohol and exercise for 48 h prior to the study visit. Water will be permitted up to 30 minutes before the study visit. Prior to initiation of study visit activities, participants will submit their 3-day food record(s) and fecal samples (if appropriate) and will be asked to complete a questionnaire detailing information about their diet, lifestyle habits, and any health issues to report. Participants will be invited to ask any questions or voice any concerns about the study visit. Then, a study coordinator will take anthropometric measures including body weight, height, waist/hip circumference and blood pressure in a private area.

Then, at study visits 1 and 2, a forearm vein catheter will be inserted for repeated blood sampling by a HHNS-approved, qualified phlebotomist. Once the catheter has been inserted, a fasting blood sample (33 mL) will be taken (baseline, time point 0). Then, participants will consume a high-fat meal (whipping cream + milk, designed to provide 1 g fat/kg body weight) containing 1500 mg of acetaminophen within 30 minutes. In addition to the high-fat meal (containing 1500 mg of acetaminophen), Acute + Chronic phase participants will consume either 3 apples or no apples at their study visit 1, and will consume the opposite (i.e. 3 apples or no apples) at study visit 2. Repeated IV blood samples (6 - 27 mL each) will be collected every 20 minutes during the first 3 hours, and then each hour for the next 3 hours, for a total of 13 blood samples (150 mL total) at each of study visits 1 and 2. Participants will be asked to remain seated for the duration of each study visit with only short walks permitted to use the washroom. Participants will be supervised by a study coordinator and/or a medically trained technician at all times throughout the study and will never be left unsupervised. After the 6-hour post-prandial period, participants will be provided with a lunch consisting of a SUBWAY sub and a juice box. Participants will be advised to avoid acetaminophen-containing products for the remainder of the day to avoid over-consumption. Total time per study visit 1 and 2 will be approximately 7 hours.

Finally, study visit 3 will conclude the Chronic phase of the study as described below.

Relevant to the Chronic phase:

Participants will visit the HNRU after a 10-12 h overnight fast on day 1 after the 2-week run-in period. Participants will be asked to consume a standardized evening meal consisting of a frozen vegetable lasagna, granola bar, pudding cup, and juice box prior to the 10-12 h overnight fast, and to avoid over-the-counter acetaminophen-containing products for 24 h, and alcohol and exercise for 48 h prior to the study visit. Water will be permitted up to 30 minutes before the study visit. Prior to initiation of study visit activities, participants will submit their 3-day food record(s) and fecal samples (if appropriate) and will be asked to complete a questionnaire detailing information about their diet, lifestyle habits, and any health issues to report. Participants will be invited to ask any questions or voice any concerns about the study visit. Then, a study coordinator will take anthropometric measures including body weight, height, waist/hip circumference and blood pressure in a private area. Afterwards, a HHNS-approved, qualified phlebotomist will conduct a venipuncture according to collect a fasting blood sample (33 mL). Finally, participants will be provided with a granola bar and juice box. Total time per study visit will be approximately 1 hour.

Procedure 4 - 3-day food records:

Participants will be asked to follow our dietary guidelines during the two-week run-in period and during the study to avoid/limit consumption of polyphenol-containing foods. Participants will be asked to complete a 3-day food record according to our instructions on 3 separate occasions: before and at the end of the 2-week run-in period and within weeks 4-6 of the Chronic phase of the study. Total time to complete 3 days of a 3-day food record will be approximately 15 minutes.

Procedure 5 - Check-in visits:

During the Chronic phase of the study, participants will be asked to visit the HNRU at the end of weeks 2 and 4 to collect more apples (or not, if in the control group), have anthropometric measures (body weight, height, waist/hip circumference and blood pressure) taken by a trained study coordinator in a private area, and complete a brief questionnaire to assess compliance with the dietary guidelines as well as recent lifestyle patterns and any health issues. Total time per check-in visit will be approximately 15 minutes.

Procedure 6 - Fecal sample collection:

On 2 occasions, prior to study visit 1 and prior to their final study visit, participants will be asked to collect 3 consecutive fecal samples according to the instructions and using the materials provided. Total time for each fecal sample collection will be approximately 5 minutes.

Procedure 7 - Study exit questionnaire:

Participants will be asked to complete a study exit questionnaire, either in-person at their final study visit or by email if the participant chooses to withdraw from the study early. Total time to complete the study exit questionnaire will be approximately 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old
* BMI ≥ 25 kg/m2 and/or waist circumference ≥ 40" for males or ≥ 30" for females
* Current/prior use of acetaminophen without complications

Exclusion Criteria:

* Pregnant or breastfeeding females
* Fasting blood glucose ≥ 7.0 mmol/L
* Chronic diseases, including by not limited to: type 2 diabetes, cardiovascular disease, liver disease, etc.
* Gastrointestinal conditions or illnesses, including but not limited to: lactose intolerance, Celiac disease, Crohn's disease, Ulcerative Colitis, Irritable Bowel Disorder
* Inflammatory conditions or active infection
* Serious major medical condition requiring hospitalization within the last year
* Taking any prescription medications (including hormonal contraceptives) or over the counter medications prescribed by a medical professional
* Taking any natural health products or dietary supplements, other than a multivitamin low in phenolic acids
* Taking any medication or natural health product contraindicated with acetaminophen
* Allergy to acetaminophen
* Use of immunomodulating agents
* Antibiotic use within last 3 months
* Alcohol consumption of ≥ 4 drinks/sitting or ≥ 14 drinks/week
* Use of tobacco products or recreational drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Plasma triglyceride levels | Fasting, and for the Acute phase of the study only: 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially
Plasma inflammatory cytokine levels | Fasting, and for the Acute phase of the study only: 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially
  E.g. adiponectin, leptin, IL-1B, IL-6, IL-10, TNF-a, MCP-1, MIP-1a, etc.
Gut microbiota profile | Immediately before and after the 6-week Chronic phase of the study
  16S rRNA gene sequencing to identify different microbes within fecal samples, representative of the gut microenvironment

SECONDARY OUTCOMES:
Fatty acid composition of chylomicron-rich fraction of blood | For the Acute phase of the study only: fasting and 120, 240, and 360 minutes post-prandially
Plasma ApoB48 levels | For the Acute phase of the study only: fasting and 120, 240, and 360 minutes post-prandially
Rate of gastric emptying | For the Acute phase of the study only: fasting and 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially
  Rate that acetaminophen (contained in the high-fat meal) appears in the blood post-prandially
Levels of inflammatory cytokines secreted from peripheral blood mononuclear cells isolated from whole blood samples and stimulated with or without lipopolysaccharide | Fasting, and for the Acute phase of the study only: 240 post-prandially
  E.g. adiponectin, leptin, IL-1B, IL-6, IL-10, TNF-a, MCP-1, MIP-1a, etc.
Plasma lipopolysaccharide binding protein | Fasting, and for the Acute phase of the study only: 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially
Plasma glucose levels | Fasting, and for the Acute phase of the study only: 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially
Plasma insulin levels | Fasting, and for the Acute phase of the study only: 20, 40, 60, 80, 100, 120, 140, 160, 180, 240, 300, and 360 minutes post-prandially

CONTACTS AND LOCATIONS:
Overall Officials: Danyelle M Liddle, MSc, Study Director — University of Guelph; Xinjie Lin, MSc, Study Director — University of Guelph
Locations (1):
- Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liddle DM , Lin X , Ward EM , Cox LC , Wright AJ , Robinson LE . Apple consumption reduces markers of postprandial inflammation following a high fat meal in overweight and obese adults: A randomized, crossover trial. Food Funct. 2021 Jul 21;12(14):6348-6362. doi: 10.1039/d1fo00392e. Epub 2021 Jun 8. PMID 34105575
- [Derived] Liddle DM, Lin X, Cox LC, Ward EM, Ansari R, Wright AJ, Robinson LE. Daily apple consumption reduces plasma and peripheral blood mononuclear cell-secreted inflammatory biomarkers in adults with overweight and obesity: a 6-week randomized, controlled, parallel-arm trial. Am J Clin Nutr. 2021 Aug 2;114(2):752-763. doi: 10.1093/ajcn/nqab094. PMID 33964852